CLINICAL TRIAL: NCT05614765
Title: Real World Data Observational Study to Evaluate the Management Status of Dyslipidemia Following Administration of Statin and Ezetimibe Complex Treatment Patient in the Medical Situation by Classification of Medical Institutions in KOREA
Brief Title: Evaluation of Dyslipidemia Management After Statin and Ezetimibe Complex Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWLC_RWE02
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: statin+ezetimibe compound
  Interventions: Drug: Statin+Ezetimibe compound

INTERVENTIONS:
Drug: Statin+Ezetimibe compound — Crezet Tablet, Litorvazet Tablet

SUMMARY:
This study is a large-scale, prospective, multi-site, and non-interventional observational study to observe the change and safety of dyslipidemia management status when administering statin+etimib complex drugs in patients with dyslipidemia.

DETAILED DESCRIPTION:
All treatments, including drug administration and laboratory tests performed after administration of statin+etimib complex, are performed by the researcher's medical judgment regardless of the subject's participation in the study, and the information to be confirmed in this observational study is collected up to 24 weeks.

Data collection will begin after the date of signing the research contract, and the follow-up period for each study subject is from the registration date (Visit 1) to the 24th week (Visit 3).

To evaluate subjects' clinical performance in real world, we collect demographic information and medical treatment based on patient's medical records, previous dyslipidemia drug administration information, blood lipid tests and liver function tests conducted at the start date of statin+etimib compound administration and subsequent 24 weeks (± 8 weeks). In the case of safety-related information, such as abnormal cases, data shall be collected at any time during the 24-week follow-up period if there is a visit by the study subject according to daily treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 19 or older as of the time of the registered visit (Visit 1)
2. Patients with dyslipidemia who are planning to administer statin+ezetimib complex or who are administering dyslipidemia complex according to the researcher's medical judgment based on the permission of statin+ezetimib complex
3. A person who can understand the information provided to him or her and voluntarily sign a written consent form

Exclusion Criteria:

1. Patients who overreact to the main ingredients or components of the drug in the study
2. Patients with active liver disease or patients with continuously high serum aminotransferase levels with unknown cause
3. Patients with muscle disease.
4. Pregnant women or pregnant women and nursing mothers
5. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabortion
6. A person who is not permitted by administration of statin+etimib complex or who falls under prohibition of administration
7. In addition to the above, a person who has determined that the researcher is not suitable for participation in this observation study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to assume the amount of LDL-C change at 24 weeks compared to the base value, the clinical trial results of the test subjects with similar underlying diseases that can be currently referred to were used.
Sampling Method: Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate and amount of change in LDL-C (measured LDL-C and calculated LDL-C) | 24 weeks
  Rate and amount of change in LDL-C (measured LDL-C and calculated LDL-C) at 24 weeks compared to baseline

SECONDARY OUTCOMES:
LDL-C change rate and amount | 12 weeks
  LDL-C change rate and amount at 12 weeks compared to baseline
Rate and amount of change in lipid variables (Non-HDL-C, HDL-C, TG, TC) | 12 weeks
  Rate and amount of change in lipid variables (Non-HDL-C, HDL-C, TG, TC) at 12 weeks compared to baseline
Rate and amount of change in lipid variables (Non-HDL-C, HDL-C, TG, TC) | 24 weeks
  Rate and amount of change in lipid variables (Non-HDL-C, HDL-C, TG, TC) at 24 weeks compared to baseline
Changes in ALT (Alanine Transaminase), AST (Aspartate Transaminase), and e-GFR (Estimated Glomerular Filtration Rate) | 12 weeks
  Changes in ALT (Alanine Transaminase), AST (Aspartate Transaminase), and e-GFR (Estimated Glomerular Filtration Rate) at 12 weeks compared to baseline
Changes in ALT (Alanine Transaminase), AST (Aspartate Transaminase), and e-GFR (Estimated Glomerular Filtration Rate) | 24 weeks
  Changes in ALT (Alanine Transaminase), AST (Aspartate Transaminase), and e-GFR (Estimated Glomerular Filtration Rate) at 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: JinWon Kim, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Not Yet decided